CLINICAL TRIAL: NCT07375316
Title: A ctDNA-guided Phase II Trial of Osimertinib in Combination With Sacituzumab Tirumotecan in EGFR-mutated Advanced NSCLC Patients With Positvie ctDNA After lead-in Osimertinib Monotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG2509
Record Dates: First submitted 2026-01-06; First posted 2026-01-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: （experimental cohort）Osimertinib + Sacituzumab Tirumotecan (Experimental): Drug: Osimertinib/Sacituzumab Tirumotecan. Osimertinib (80mg QD) + Sacituzumab Tirumotecan (4 mg/m2) on Day 1 and Day 8 of 28-day cycles (4 mg/m2 Q2W).
  Interventions: Drug: Osimertinib + Sacituzumab Tirumotecan
- Cohort 2: （observational cohort）Osimertinib monotherapy (Active Comparator): Drug: Osimertinib •Osimertinib (80mg QD).
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib + Sacituzumab Tirumotecan — Osimertinib (80mg QD) + Sacituzumab Tirumotecan (4 mg/m2) on Day 1 and Day 8 of 28-day cycles (4 mg/m2 Q2W).
  Arms: Cohort 1: （experimental cohort）Osimertinib + Sacituzumab Tirumotecan
Drug: Osimertinib — Osimertinib (80mg QD)
  Arms: Cohort 2: （observational cohort）Osimertinib monotherapy

SUMMARY:
EGFR-mutated advanced NSCLC patients without ctDNA clearance after lead-in osimertinib monotherapy have inferior PFS compared with those with ctDNA clearance. Consequently, these patients might need an intensified therapeutic strategy, such as osimertinib combined with chemotherapy or ADC. This study aims to explore the efficacy and safety of osimertinib in combination with sacituzumab tirumotecan adaptively in EGFR-mutated advanced NSCLC patients with positive ctDNA after lead-in osimertinib monotherapy.

DETAILED DESCRIPTION:
This is an investigator-initiated, multicenter, ctDNA-guided phase II study to evaluate the efficacy and safety of osimertinib in combination with sacituzumab tirumotecan adaptively in EGFR-mutated advanced NSCLC patients with positive ctDNA after lead-in osimertinib monotherapy (Cohort 1). Patients screened to be with negative ctDNA after lead-in osimertinib will be prospectively enrolled in a real-world cohort to observe PFS on continued osimertinib monotherapy (Cohort 2).

Approximately 120 eligible patients are planned to undergo tumor assessment and ctDNA testing upon completion of one cycle (3 weeks per cycle) treatment with osimertinib (obtained commercially at the standard dose of 80mg orally daily). Patients without disease progression assessed by imaging will be enrolled into different study cohorts based on ctDNA test results.

Only patients who test positive for ctDNA will be enrolled in Cohort 1 of the clinical study to receive the combinational treatment of intravenous sac-TMT at a fixed dose of 4mg/kg every 2 weeks plus oral osimertinib also at a fixed dose of 80mg daily until disease progression, death, unacceptable toxicity, or another treatment discontinuation criterion is met, whichever occurs first.

Patients who test negative for ctDNA will continue to receive osimertinib monotherapy and be prospectively enrolled in observational Cohort 2. In this observational cohort, treatments and treatment-related data collection are at the discretion of physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of signing the Informed Consent Form (ICF), regardless of gender;
2. Histologically or cytologically confirmed locally advanced (stage IIIB/IIIC) or metastatic (Stage IV) non-squamous NSCLC not amenable to radical surgery and/or radical radiotherapy (regardless of concurrent/sequential chemotherapy) (according to TNM staging of lung cancer published by the Union for International Cancer Control and American Joint Committee on Cancer (UICC/AJCC), 8th edition);
3. Presence of sensitizing EGFR mutation (exon 19 deletion and/or L858R);
4. Completion of 3-week first-line treatment with osimertinib monotherapy. Non-PD as assessed by investigator per RECIST v1.1, and willing to undergo ctDNA testing (patients with positive ctDNA test results will be enrolled in Cohort 1; patients with negative ctDNA test results will be enrolled in observational Cohort 2);
5. ≥1 measurable target lesion per RECIST v1.1;
6. ECOG Performance Status score of 0 or 1 within 7 days before enrollment;
7. Adequate organ and bone marrow function (no blood transfusion, recombinant human thrombopoietin, or colony stimulating factor therapy within 2 weeks prior to the first dose), defined as follows:

   1. Hematology: neutrophil count (NEUT) ≥ 1.5×109/L; platelet (PLT) ≥ 100×109/L; hemoglobin(Hb) ≥ 90g/L;
   2. Liver function: AST and ALT ≤ 2.5× ULN (if liver metastases are present, ≤5 × ULN); total bilirubin (TBIL) ≤ 1.5×ULN (if liver metastases are present, ≤3 × ULN); serum albumin ≥30g/L;
   3. Renal function: serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min (calculated using the standard Cockcroft-Gault formula);
   4. Coagulation function: international normalized ratio (INR), activated partial thromboplastin time (APTT) and prothrombin time (PT) ≤ 1.5× ULN;
8. Use of effective medical contraception during the study treatment period and for 6 months after the end of dosing for female subjects of childbearing potential and male subjects with partners of childbearing potential;
9. Willingness to participate in the study, sign the ICF, and comply with the protocol-specified visits and relevant procedures.

Exclusion Criteria:

1. For NSCLC, histologically or cytologically confirmed squamous cell carcinoma component or presence of coexisting small cell lung cancer, neuroendocrine carcinoma, or carcinosarcoma component;
2. Known presence of meningeal metastases, brainstem metastases, spinal cord metastases and/or compression, and active brain metastases;
3. Prior treatment with systemic anti-tumor therapy for locally advanced or metastatic NSCLC other than osimertinib;
4. Prior treatment with any TROP2-targeted therapy or any therapy that targets topoisomerase I (including ADCs);
5. Other malignancies (except cured local tumors, such as basal cell carcinoma of skin, squamous cell carcinoma of skin, carcinoma in situ of the cervix) within 3 years prior to enrollment;
6. Presence of any of the following cardiovascular and cerebrovascular diseases or risk factors:

   1. Myocardial infarction, unstable angina, acute or persistent myocardial ischemia, Class III or IV heart failure [according to New York Heart Association (NYHA) classification], symptomatic or poorly controlled serious arrhythmia, cerebrovascular accident, transient ischemic attack, and other serious cardiovascular and cerebrovascular diseases within 6 months prior to enrollment;
   2. Previous history of myocardial diseases such as myocarditis, primary cardiomyopathy and specific cardiomyopathy;
   3. Any peripheral arterial thromboembolic event, pulmonary embolism, deep vein thrombosis, or other serious thromboembolic event within 3 months prior to enrollment;
   4. Major vascular disease such as aortic aneurysm, aortic dissecting aneurysm that may be life-threatening or require surgery within 6 months prior to first dose;
   5. Mean corrected QT interval (QTcF) between ventricular depolarization to repolarization > 470 ms;
7. Uncontrolled systemic disease as judged by the investigator:

   1. Poorly controlled diabetes mellitus (two consecutive fasting glucose ≥10 mmol/L);
   2. Poorly controlled hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg);
   3. Presence of clinically symptomatic pleural effusion, pericardial effusion, or ascites requiring repeated drainage (> 1 time/week);
8. History of (noninfectious) pneumonitis/interstitial lung disease (ILD) that required steroids, or has current pneumonitis/ILD, or suspected pneumonitis/ILD that cannot be ruled out by imaging at screening;
9. Documented severe dry eye syndrome, severe meibomian gland disease and/or blepharitis, or history of corneal disease that prevents/delays corneal healing;
10. Clinically severe lung impairment caused by complications that may involve the lung, or prior pneumonectomy;
11. Presence of active chronic inflammatory bowel disease, GI tract obstruction, severe ulcers, gastrointestinal perforation, abdominal abscess, or acute GI tract bleed;
12. Active gastrointestinal disease or other conditions that significantly affect the absorption and metabolism of osimertinib (e.g., refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow drug, or previous major bowel resection);
13. Tumor invasion or compression of surrounding important organs and blood vessels (e.g. heart, esophagus, superior vena cava, etc.) accompanied by related symptoms (e.g. superior vena cava syndrome), or presence of risk of developing esophagotracheal fistula or esophagopleural fistula;
14. Toxicities treated by prior anti-tumor therapy having not recovered to ≤ Grade 1 (as per NCI CTCAE V5.0) or to the levels specified in the eligibility criteria;
15. Serious infection within 4 weeks prior to enrollment or active infection requiring systemic anti-infective therapy within 2 weeks prior to enrollment;
16. Known active tuberculosis;
17. Presence of active hepatitis B (HBV-DNA test is required in case of hepatitis B surface antigen [HBsAg] positive; HBV-DNA ≥ 500 IU/mL or above the lower limit of detection, whichever is higher) or hepatitis C (hepatitis C antibody positive, and HCV-RNA > the lower limit of detection);
18. Positive result of human immunodeficiency virus (HIV) test or history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection;
19. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
20. Major surgery within 4 weeks prior to enrollment or expected major surgery during the study;
21. Known allergy to the study drug or any of its components, and a history of known severe hypersensitivity to other monoclonal antibodies;
22. Medications or herbal supplements that are currently used (or cannot be discontinued prior to receiving the first dose of study treatment) and are known to be strong inducers or inhibitors of cytochrome P450 (CYP) 3A4 (washout for at least 3 weeks);
23. Receipt of radiotherapy at a total dose of >30 Gy for lung lesions within 6 months prior to enrollment; receipt of non-thoracic or extensive radiotherapy at a total dose of >30 Gy within 4 weeks prior to enrollment; palliative radiotherapy for symptom control is allowed, but must be completed at least 2 weeks prior to enrollment;
24. Live vaccines inoculated within 30 days prior to enrollment or planned to be inoculated during the study;
25. Rapid deterioration of disease, such as significant changes in performance status during the screening process prior to the first dose;
26. Pregnant or lactating women;
27. Any condition that, in the opinion of the investigator, may interfere with the evaluation of the study drug or the interpretation of the subject's safety or study results, or any other circumstances that, in the opinion of the investigator, make the subject unsuitable for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) in Cohort 1, Assessed by Investigator | From date of start of combinational treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  PFS is defined as time from the date of start of combinational treatment until the date of disease progression per RECIST 1.1, as assessed by investigator, or death due to any cause.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) in Cohort 1, Assessed by Investigator | Tumour assessments will be conducted according to the RECIST v1.1, with valuations performed every six weeks during the first year after first dose and every 12 weeks thereafter, up to 36 months.
  ORR is defined as the percentage of subjects who have a best overall response of Complete Response (CR) or Partial Response (PR) per RECIST 1.1 as assessed by the Investigator.
Disease Control Rate (DCR) in Cohort 1, Assessed by Investigator | Tumour assessments will be conducted according to the RECIST v1.1, with valuations performed every six weeks during the first year after first dose and every 12 weeks thereafter, up to 36 months.
  DCR is defined as the percentage of subjects who have a best overall response of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) per RECIST 1.1 as assessed by the Investigator.
Overall Survival (OS) in Cohort 1 | From date of start of combinational treatment until the date of death from any cause, assessed up to 36 months
  OS is defined as the time from the date of start of combinational treatment until the date of death due to any cause.
Adverse Events in Cohort 1 | From the start of study drug to 30 days after the last dose of study drug
  The number of patients with adverse events and the severity according to CTCAE v5.0.
Progression-free survival in Cohort 2, Assessed by Investigator | From date of start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  PFS is defined as time from the date of start of treatment until the date of disease progression per RECIST 1.1, as assessed by investigator, or death due to any cause.

OTHER OUTCOMES:
Biomarkers in Cohort 1 | The data of ctDNA clearance rate will be collected at 2 time points: at the completion of induction treatment with osimertinib, and 6 weeks after first dose of study treatment.
  The proportion of patients with circulating tumor DNA clearance after 6 weeks study treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Guangdong Lung Cancer Institute, Guangdong Provincial People's Hospital (Guangdong Academy of Medical Sciences), Southern Medical University, Guangzhou, Guangdong
  - Meizhou People's Hospital (Huangtang Hospital), Meizhou Academy of Medical Sciences, Meizhou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No